CLINICAL TRIAL: NCT05088226
Title: Ruxolitinib and Chidamide Intensified Bu/CY Conditioning Regimen for Patients With Acute B Cell Lymphoblast Leukemia Underwenting Haploidenticl Peripheral Blood Stem Cell Transplantation
Brief Title: Ruxolitinib and Chidamide Intensified Bu/CY Conditioning Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2020-483-01
Record Dates: First submitted 2021-05-25; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Blood Stem Cell Transplantation
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib combined with Chidamide (Experimental): Experimental: Ruxolitinib combined with Chidamide. All recipients in this arm received the modified Bu/Cy conditioning regimen intensified by Ruxolitinib and Chidamide. The conditioning regimen for allogeneic hematopoietic stem cell transplantation consist of ruxolitinib (35 mg bid [p.o.], days -15 to -10, diminishing to day -1), chidamide (30 mg/day, twice per week from days -15 to -2), cytarabine (4g/m2/day, days -10 to -9), busulfan (0.8mg/kg, Q6h, days -8 to -6), cyclophosphamide (1.8 g/m2/day, days -5 to -4), carmustine(BCNU) (250mg/m2/day, day -3)
  Interventions: Drug: Ruxolitinib combined with Chidamide.

INTERVENTIONS:
Drug: Ruxolitinib combined with Chidamide. — Drug: modified By/Cy conditioning regimen intensified by Ruxolitinib and Chidamide .
  Day -15 # Ruxolitinib 70mg bid, Chidamide 30 mg once; Day -14 # Ruxolitinib 70mg bid; Day -13 # Ruxolitinib 70mg bid; Day -12 # Ruxolitinib 70mg bid, Chidamide 30 mg once; Day -11 # Ruxolitinib 70mg bid; Day-10# Cytarabine 4g/m2/day CI , Ruxolitinib 60mg bid; Day- 9# Cytarabine 4g/m2/day CI, Ruxolitinib 60mg bid; Day- 8 # Busulfan 0.8mg/ kg Q6h iv, Ruxolitinib 50mg bid, Chidamide 30 mg once; Day- 7# Busulfan 0.8mg/ kg Q6h iv, Ruxolitinib 50mg bid; Day-6# Busulfan 0.8mg/kg Q6h iv, Ruxolitinib 40mg bid; Day-5# Cyclophosphamide 1.8 g/m2/day CI, Ruxolitinib 30mg bid, Chidamide 30 mg once; Day-4# Cyclophosphamide 1.8 g/m2/day CI,Ruxolitinib 20mg bid; Day-3# Carmustine 250mg/m2/ day iv, Ruxolitinib 10mg bid; Day-2# Ruxolitinib 5mg bid, Chidamide 30 mg/day; Day-1# Ruxolitinib 5mg qd;
  Other Names: Modified By/Cy conditioning regimen intensified by Ruxolitinib and Chidamide

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Ruxolitinib and Chidamide intensified conditioning regimen in patients with Acute B cell Lymphoblast leukemia Underwenting Haploidenticl Peripheral blood Stem Cell Transplantation.

DETAILED DESCRIPTION:
Haploidenticl Peripheral blood Stem Cell Transplantation should be offered to eligible patients with Acute B cell Lymphoblast leukemia whenever feasible. To further improve the outcome of transplantation patients with Acute B cell Lymphoblast leukemia, we developed a modified Bu/Cy conditioning regimen intensified by Ruxolitinib and Chidamide. In this study, we tested the efficacy and feasibility of the modified Bu/Cy conditioning regimen intensified by Ruxolitinib and Chidamide in patients with Acute B cell Lymphoblast leukemia undergoing allogeneic peripheral blood stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. high risk acute B cell lymphoblastic leukemia with the indications for allogeneic transplantation;
2. Have matched sibling donors, ≥8/10 HLA matched unrelated donors or haploidentical donors
3. All patients should aged 12 to 65 years;
4. Liver function: ALT and AST≤2.5 times the upper limit of normal , bilirubin≤2 times the upper limit of normal;
5. Renal function: creatinine ≤the upper limit of normal;
6. Patients without any uncontrolled infections , without organ dysfunction or without severe mental illness;
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
8. Have signed informed consent.

Exclusion Criteria:

1. pregnant women;
2. Patients with mental illness or other states unable to comply with the protocol;
3. ALL patients with Ph positive;

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants relapse as assessed by NCCN (National Comprehensive Cancer Network ) criteria | 365 days after transplantation
  Defined as the proportion of participants whose underlying malignancy relapsed.

SECONDARY OUTCOMES:
DFS(disease-free survival ) | 365 days after transplantation
  DFS was defined as survival with no evidence of relapse or progression.
TRM(treatment-related mortality ) | 365 days after transplantation
  Defined as the proportion of subjects who died due to causes other than malignancy relapse.
Proportion of participants with aGVHD as assessed by acute graft versus host disease grading criteria (refer to Glucksberg criteria) | 365 days after transplantation
  Defined as the proportion of participants who developed acute GVHD.
Proportion of participants with cGVHD as assessed by chronic graft versus host disease grading criteria (refer to NIH criteria) | 365 days after transplantation
  Defined as the proportion of participants who developed chronic GVHD.
OS(overall survival ) | 365 days after transplantation
  OS was defined as the time from transplantation to death due to any cause.
Failure-free survival (FFS) | 365 days after transplantation
  Defined as the time from tranplantation to the earliest date that a participant died, had a relapse/progression of the underlying malignancy, required additional therapy for aGVHD, or demonstrated signs or symptoms of chronic graft-versus-host disease (cGVHD).
infection rate | 365 days after transplantation
  Defined as the proportion of participants who developed all kinds of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maude SL, Dolai S, Delgado-Martin C, Vincent T, Robbins A, Selvanathan A, Ryan T, Hall J, Wood AC, Tasian SK, Hunger SP, Loh ML, Mullighan CG, Wood BL, Hermiston ML, Grupp SA, Lock RB, Teachey DT. Efficacy of JAK/STAT pathway inhibition in murine xenograft models of early T-cell precursor (ETP) acute lymphoblastic leukemia. Blood. 2015 Mar 12;125(11):1759-67. doi: 10.1182/blood-2014-06-580480. Epub 2015 Feb 2. PMID 25645356
- [Background] Delgado-Martin C, Meyer LK, Huang BJ, Shimano KA, Zinter MS, Nguyen JV, Smith GA, Taunton J, Winter SS, Roderick JR, Kelliher MA, Horton TM, Wood BL, Teachey DT, Hermiston ML. JAK/STAT pathway inhibition overcomes IL7-induced glucocorticoid resistance in a subset of human T-cell acute lymphoblastic leukemias. Leukemia. 2017 Dec;31(12):2568-2576. doi: 10.1038/leu.2017.136. Epub 2017 May 9. PMID 28484265
- [Background] Shi Y, Jia B, Xu W, Li W, Liu T, Liu P, Zhao W, Zhang H, Sun X, Yang H, Zhang X, Jin J, Jin Z, Li Z, Qiu L, Dong M, Huang X, Luo Y, Wang X, Wang X, Wu J, Xu J, Yi P, Zhou J, He H, Liu L, Shen J, Tang X, Wang J, Yang J, Zeng Q, Zhang Z, Cai Z, Chen X, Ding K, Hou M, Huang H, Li X, Liang R, Liu Q, Song Y, Su H, Gao Y, Liu L, Luo J, Su L, Sun Z, Tan H, Wang H, Wang J, Wang S, Zhang H, Zhang X, Zhou D, Bai O, Wu G, Zhang L, Zhang Y. Chidamide in relapsed or refractory peripheral T cell lymphoma: a multicenter real-world study in China. J Hematol Oncol. 2017 Mar 15;10(1):69. doi: 10.1186/s13045-017-0439-6. PMID 28298231
- [Background] Savino AM, Sarno J, Trentin L, Vieri M, Fazio G, Bardini M, Bugarin C, Fossati G, Davis KL, Gaipa G, Izraeli S, Meyer LH, Nolan GP, Biondi A, Te Kronnie G, Palmi C, Cazzaniga G. The histone deacetylase inhibitor givinostat (ITF2357) exhibits potent anti-tumor activity against CRLF2-rearranged BCP-ALL. Leukemia. 2017 Nov;31(11):2365-2375. doi: 10.1038/leu.2017.93. Epub 2017 Mar 23. PMID 28331226
- [Background] Ding YY, Stern JW, Jubelirer TF, Wertheim GB, Lin F, Chang F, Gu Z, Mullighan CG, Li Y, Harvey RC, Chen IM, Willman CL, Hunger SP, Li MM, Tasian SK. Clinical efficacy of ruxolitinib and chemotherapy in a child with Philadelphia chromosome-like acute lymphoblastic leukemia with GOLGA5-JAK2 fusion and induction failure. Haematologica. 2018 Sep;103(9):e427-e431. doi: 10.3324/haematol.2018.192088. Epub 2018 May 17. No abstract available. PMID 29773603
- [Background] Ferrante F, Giaimo BD, Bartkuhn M, Zimmermann T, Close V, Mertens D, Nist A, Stiewe T, Meier-Soelch J, Kracht M, Just S, Kloble P, Oswald F, Borggrefe T. HDAC3 functions as a positive regulator in Notch signal transduction. Nucleic Acids Res. 2020 Apr 17;48(7):3496-3512. doi: 10.1093/nar/gkaa088. PMID 32107550